CLINICAL TRIAL: NCT02925117
Title: A Phase 2b Multicenter, Randomized, Placebo-Controlled, Double-Blind Dose-Ranging Study to Evaluate ABT-494 (Upadacitinib) in Adult Subjects With Moderate to Severe Atopic Dermatitis
Brief Title: A Study to Evaluate ABT-494 (Upadacitinib) in Adults With Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-048; 2016-002451-21 (EudraCT Number)
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Results first posted 2020-07-16 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Atopic Dermatitis
Keywords: ABT-494; Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — upadacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Placebo (Placebo Comparator): Participants randomized to receive placebo once daily (QD) for 16 weeks in Period 1. At Week 16 participants were re-randomized to receive 30 mg upadacitinib or placebo once a day for 72 weeks in Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Upadacitinib 7.5 mg (Experimental): Participants randomized to receive upadacitinib 7.5 mg QD for 16 weeks in Period 1. At Week 16 participants were re-randomized to receive 7.5 mg upadacitinib or placebo QD for 72 weeks in Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Upadacitinib 15 mg (Experimental): Participants randomized to receive upadacitinib 15 mg QD for 16 weeks in Period 1. At Week 16 participants were re-randomized to receive 15 mg upadacitinib or placebo QD for 72 weeks in Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo
- Upadacitinib 30 mg (Experimental): Participants randomized to receive upadacitinib 30 mg QD for 16 weeks in Period 1. At Week 16 participants were re-randomized to receive 30 mg upadacitinib or placebo QD for 72 weeks in Period 2.
  Interventions: Drug: Upadacitinib; Drug: Placebo

INTERVENTIONS:
Drug: Upadacitinib — Tablet for oral use
  Other Names: RINVOQ™; ABT-494
Drug: Placebo — Tablet

SUMMARY:
The objective of this study was to evaluate the safety and efficacy of multiple doses of upadacitinib monotherapy versus placebo in the treatment of adults with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
The study was to include a 16-week double-blind treatment period (Period 1) and a 72-week double-blind treatment period (Period 2) for a total of 88 weeks of treatment. Participants who met eligibility criteria were to be randomized in a 1:1:1:1 ratio to one of the four treatment groups. Participants who completed Period 1 were re-randomized at Week 16 into a 72-week double-blind, placebo-controlled treatment period (Period 2) in a 1:1 ratio:

* Group 1: Upadacitinib 7.5 mg once daily (QD) (Day 1 to Week 16) → upadacitinib 7.5 mg QD or placebo (Week 16 - and thereafter)
* Group 2: Upadacitinib 15 mg QD (Day 1 to Week 16) → upadacitinib 15 mg QD or placebo (Week 16 and thereafter)
* Group 3: Upadacitinib 30 mg QD (Day 1 to Week 16) → upadacitinib 30 mg QD or placebo (Week 16 - and thereafter)
* Group 4: Matching placebo (Day 1 to Week 16) → upadacitinib 30 mg QD or placebo (Week 16 and thereafter)

In Period 1, discontinuation from study drug was mandatory for any participant with an Eczema Area and Severity Index (EASI) score worsening of 25% or more compared with their Baseline EASI score at any 2 consecutive scheduled study visits from Week 4 to Week 12.

In Period 2, blinded rescue therapy with upadacitinib 30 mg QD was provided after the first instance of a < EASI 50 response starting at the Week 20 visit (4 weeks after re-randomization into Period 2) for the remainder of the study.

ELIGIBILITY:
Inclusion Criteria:

* Atopic dermatitis with a diagnosis confirmed by a dermatologist (according to the Hanifin and Rajka criteria) and onset of symptoms at least 1 year prior to Baseline.
* Moderate to severe atopic dermatitis defined by an Eczema Area and Severity Index (EASI) ≥ 16, body surface area (BSA) ≥ 10% and an Investigators Global Assessment (IGA) score ≥ 3 at the Baseline visit.
* Documented history (within 1 year prior to the screening visit) of inadequate response to treatment with topical corticosteroids (TCS), or topical calcineurin inhibitors (TCI), or for whom topical treatments are otherwise medically inadvisable (e.g., because of important side effects or safety risks).
* Twice daily use of an additive-free, bland emollient for at least 7 days prior to Baseline.

Exclusion Criteria:

* Prior exposure to any systemic or topical Janus kinase (JAK) inhibitor (including but not limited to tofacitinib, baricitinib, ruxolitinib, and filgotinib).
* Treatment with topical corticosteroids (TCS), topical calcineurin inhibitors (TCI), prescription moisturizers or moisturizers containing additives such as ceramide, hyaluronic acid, urea, or filaggrin within 10 days prior to the Baseline visit.
* Prior exposure to dupilumab or exposure to systemic therapies for AD including corticosteroids, methotrexate, cyclosporine, azathioprine, phosphodiesterase type 4 (PDE4)-inhibitors and mycophenolate mofetil within 4 weeks prior to Baseline.
* Prior exposure to any investigational systemic treatment within 30 days or 5 half-lives (whichever is longer) of the Baseline visit or is currently enrolled in another clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2016-10-25 (Actual); Primary Completion 2017-08-10 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (34):
- United States (10):
  - ForCare Clinical Research /ID# 157974, Tampa, Florida
  - Advanced Medical Research /ID# 154516, Sandy Springs, Georgia
  - DermAssociates /ID# 153584, Rockville, Maryland
  - Tufts Medical Center /ID# 153586, Boston, Massachusetts
  - Psoriasis Treatment Ctr NJ /ID# 153578, East Windsor, New Jersey
  - Icahn School of Med Mt. Sinai /ID# 153582, New York, New York
  - Univ Rochester Med Ctr /ID# 154477, Rochester, New York
  - Arlington Research Center, Inc /ID# 154522, Arlington, Texas
  - Modern Research Associates, PL /ID# 154487, Dallas, Texas
  - Center for Clinical Studies /ID# 153589, Houston, Texas
- Australia (4):
  - Woden Dermatology /ID# 157907, Phillip, Australian Capital Territory
  - St George Hospital /ID# 157908, Kogarah, New South Wales
  - Specialist Connect Pty Ltd /ID# 157909, Woolloongabba, Queensland
  - Skin Health Institute Inc /ID# 157906, Carlton, Victoria
- Canada (7):
  - Institute for Skin Advancement /ID# 153246, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc. /ID# 153241, Surrey, British Columbia
  - Enverus Medical Research /ID# 153239, Surrey, British Columbia
  - CCA Medical Research /ID# 155817, Ajax, Ontario
  - Lynderm Research Inc. /ID# 153242, Markham, Ontario
  - Dermatology Ottawa Research Centre /ID# 153248, Ottawa, Ontario
  - K. Papp Clinical Research /ID# 153244, Waterloo, Ontario
- Finland (2):
  - Mehiläinen Neo /ID# 154960, Turku, Southwest Finland
  - Mikkeli Central Hospital /ID# 154959, Mikkeli
- TFS Trial Form Support GmbH /ID# 155442, Hamburg, Germany
- Japan (4):
  - Fukuoka University Hospital /ID# 152714, Fukuoka, Fukuoka
  - Takagi Dermatological Clinic /ID# 152706, Obihiro-shi, Hokkaido
  - Medical Cooperation Kojinkai Sapporo Skin Clinic /ID# 153781, Sapporo, Hokkaido
  - Nippon Medical School Hospital /ID# 153287, Tokyo
- Netherlands (4):
  - Radboud Universitair Medisch Centrum /ID# 153688, Nijmegen, Gelderland
  - Academisch Medisch Centrum /ID# 153596, Amsterdam, North Holland
  - Universitair Medisch Centrum Groningen /ID# 153595, Groningen
  - Universitair Medisch Centrum Utrecht /ID# 153687, Utrecht
- Spain (2):
  - Hospital Santa Creu i Sant Pau /ID# 153519, Barcelona
  - Hospital Univ Germans Trias I /ID# 155598, Barcelona

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Result] Guttman-Yassky E, Thaci D, Pangan AL, Hong HC, Papp KA, Reich K, Beck LA, Mohamed MF, Othman AA, Anderson JK, Gu Y, Teixeira HD, Silverberg JI. Upadacitinib in adults with moderate to severe atopic dermatitis: 16-week results from a randomized, placebo-controlled trial. J Allergy Clin Immunol. 2020 Mar;145(3):877-884. doi: 10.1016/j.jaci.2019.11.025. Epub 2019 Nov 29. PMID 31786154

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 36 sites in 8 countries (Australia, Canada, Finland, Germany, Japan, Netherlands, Spain, and the United States [US]).
  The study included a 16-week double-blind treatment period (Period 1) followed by a a 72-week double-blind treatment period (Period 2) for a total of 88 weeks of treatment.
Pre-assignment Details: Participants were randomized in a 1:1:1:1 ratio, stratified by geographic region (US and Canada; European Union and Australia; and Japan). Participants who completed Period 1 were re-randomized at Week 16 in a 1:1 ratio within their original treatment group assignments to either upadacitinib or placebo. Rescue therapy was provided from Week 20.
Groups:
- Placebo / Placebo: Participants originally randomized to placebo were re-randomized at Week 16 to receive placebo tablets once a day for 72 weeks in Period 2.
- Placebo / Upadacitinib 30 mg: Participants originally randomized to placebo were re-randomized at Week 16 to receive 30 mg upadacitinib once a day for 72 weeks in Period 2.
- Upadacitinib 7.5 mg / Placebo: Participants originally randomized to 7.5 mg upadacitinib were re-randomized at Week 16 to receive placebo tablets once a day for 72 weeks in Period 2.
- Upadacitinib 7.5 mg / Upadacitinib 7.5 mg: Participants originally randomized to 7.5 mg upadacitinib were re-randomized at Week 16 to receive 7.5 mg upadacitinib once a day for 72 weeks in Period 2.
- Upadacitinib 15 mg / Placebo: Participants originally randomized to 15 mg upadacitinib were re-randomized at Week 16 to receive placebo tablets once a day for 72 weeks in Period 2.
- Upadacitinib 15 mg / Upadacitinib 15 mg: Participants originally randomized to 15 mg upadacitinib were re-randomized at Week 16 to receive 15 mg upadacitinib once a day for 72 weeks in Period 2.
- Upadacitinib 30 mg / Placebo: Participants originally randomized to 30 mg upadacitinib were re-randomized at Week 16 to receive placebo tablets once a day for 72 weeks in Period 2.
- Upadacitinib 30 mg / Upadacitinib 30 mg: Participants originally randomized to 30 mg upadacitinib were re-randomized at Week 16 to receive 30 mg upadacitinib once a day for 72 weeks in Period 2.
Period: Period 1 (Weeks 0 - 16)
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Placebo / Placebo | Placebo / Upadacitinib 30 mg | Upadacitinib 7.5 mg / Placebo | Upadacitinib 7.5 mg / Upadacitinib 7.5 mg | Upadacitinib 15 mg / Placebo | Upadacitinib 15 mg / Upadacitinib 15 mg | Upadacitinib 30 mg / Placebo | Upadacitinib 30 mg / Upadacitinib 30 mg
Started | 41 | 42 | 42 | 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received Treatment | 40 | 42 | 42 | 42 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 23 | 31 | 37 | 39 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 18 | 11 | 5 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 3 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 4 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 2 (Weeks 16 - 88)
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Placebo / Placebo | Placebo / Upadacitinib 30 mg | Upadacitinib 7.5 mg / Placebo | Upadacitinib 7.5 mg / Upadacitinib 7.5 mg | Upadacitinib 15 mg / Placebo | Upadacitinib 15 mg / Upadacitinib 15 mg | Upadacitinib 30 mg / Placebo | Upadacitinib 30 mg / Upadacitinib 30 mg
Started (Four participants completed Week 16 but were not re-randomized into Period 2.) | 0 | 0 | 0 | 0 | 10 | 10 | 15 | 16 | 19 | 18 | 19 | 19
Rescued to Upadacitinib 30 mg | 0 | 0 | 0 | 0 | 8 | 1 | 13 | 12 | 17 | 12 | 14 | 4
Completed | 0 | 0 | 0 | 0 | 8 | 5 | 9 | 11 | 13 | 12 | 11 | 14
Not Completed | 0 | 0 | 0 | 0 | 2 | 5 | 6 | 5 | 6 | 6 | 8 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 4 | 3 | 2 | 2 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 1 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 3 | 4 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants (intent-to-treat population)
Groups:
- Placebo: Participants randomized to receive placebo once daily (QD) for 16 weeks in Period 1.
- Upadacitinib 7.5 mg: Participants randomized to receive upadacitinib 7.5 mg QD for 16 weeks in Period 1.
- Upadacitinib 15 mg: Participants randomized to receive upadacitinib 15 mg QD for 16 weeks in Period 1.
- Upadacitinib 30 mg: Participants randomized to receive upadacitinib 30 mg QD for 16 weeks in Period 1.
- Total: Total of all reporting groups
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg | Total
Number analyzed (Participants) | 41 | 42 | 42 | 42 | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (17.52) | 41.5 (15.36) | 38.5 (15.24) | 39.9 (15.30) | 39.9 (15.77)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 25 | 22 | 25 | 22 | 94
  40 - 64 years | 11 | 16 | 14 | 17 | 58
  ≥ 65 years | 5 | 4 | 3 | 3 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 12 | 20 | 63
  Male | 24 | 28 | 30 | 22 | 104
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 41 | 40 | 40 | 41 | 162
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 24 | 21 | 23 | 96
  Black or African American | 6 | 7 | 10 | 6 | 29
  Asian | 7 | 9 | 9 | 13 | 38
  American Indian/Alaska Native | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 1 | 0 | 3
Geographic Region [Count of Participants; unit: Participants]
  US/Canada | 29 | 29 | 29 | 29 | 116
  EU/Australia | 10 | 11 | 10 | 10 | 41
  Japan | 2 | 2 | 3 | 3 | 10
Duration of Atopic Dermatitis Diagnosis [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 40 | 42 | 42 | 42 | 166
    (all) | 26.84 (18.76) | 30.44 (18.07) | 22.59 (15.78) | 24.24 (13.58) | 26.02 (16.76)
Eczema Area and Severity Index (EASI) [Mean (Standard Deviation); unit: units on a scale] — EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  units on a scale | 32.62 (14.49) | 31.42 (15.76) | 31.40 (12.26) | 28.15 (11.62) | 30.89 (13.61)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Eczema Area and Severity Index (EASI) Score at Week 16
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1], moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from baseline indicates improvement.
Time Frame: Baseline and Week 16
Population: Randomized participants with at least one post-baseline EASI assessment; last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 39 | 42 | 42 | 42
percent change | -23.0 (6.42) | -39.4 (6.24) | -61.7 (6.12) | -74.4 (6.13)
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) with stratum (geographic region), baseline value, and treatment in the model; Least Squares (LS) Mean Difference = -51.4, 95% CI 2-sided [-66.5 to -36.3], Standard Error of Mean 7.65
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; Analysis of covariance (ANCOVA) with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -38.7, 95% CI 2-sided [-53.7 to -23.6], Standard Error of Mean 7.61
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.032, ANCOVA; Analysis of covariance (ANCOVA) with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -16.4, 95% CI 2-sided [-31.4 to -1.4], Standard Error of Mean 7.61

2. Secondary Outcome: Percentage of Participants Who Achieved a 75% Reduction in EASI Score (EASI 75) at Week 16
Description: EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  An EASI 75 response is defined as participants with at least a 75% reduction (improvement) in EASI score relative to the Baseline value.
  Participants with missing values at Week 16 were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Week 16
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants | 9.8 | 28.6 | 52.4 | 69.0
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, adjusted for stratum (geographic region); Adjusted Difference = 58.7, 95% CI 2-sided [42.5 to 74.8]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, adjusted for stratum (geographic region); Adjusted Difference = 42.5, 95% CI 2-sided [25.5 to 59.6]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.022, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, adjusted for stratum (geographic region); Adjusted Difference = 18.7, 95% CI 2-sided [2.7 to 34.7]

3. Secondary Outcome: Percentage of Participants Achieving an Investigator Global Assessment (IGA) of "0" or "1" at Week 16
Description: The Investigator's Global Assessment for Atopic Dermatitis (IGA) was scored on the following scale:
  * 0: Clear (No inflammatory signs of atopic dermatitis)
  * 1: Almost Clear (Just perceptible erythema and just perceptible papulation/infiltration)
  * 2: Mild (Mild erythema and mild papulation/infiltration)
  * 3: Moderate (Moderate erythema and moderate papulation/infiltration)
  * 4: Severe (Severe erythema and severe papulation/infiltration with or without oozing/crusting)
  The percentage of participants with a score of 0 or 1 at Week 16 is reported.
Time Frame: Week 16
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants | 2.4 | 14.3 | 31.0 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, adjusted for stratum (geographic region); Adjusted Difference = 46.9, 95% CI 2-sided [31.1 to 62.7]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, adjusted for stratum (geographic region); Adjusted Difference = 28.6, 95% CI 2-sided [13.8 to 43.4]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.044, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test, adjusted for stratum (geographic region); Adjusted Difference = 11.9, 95% CI 2-sided [0.3 to 23.5]

4. Secondary Outcome: Percent Change From Baseline to Weeks 2, 8, and 16 in Pruritus Numerical Rating Scale (NRS)
Description: Participants were asked to rate pruritus (itch) in the past 24 hours on a daily basis using a scale from 0 to 10, with 0 being no itch and 10 being the worst imaginable itch. The percent change from Baseline at each week was calculated from a rolling weekly average.
Time Frame: Baseline and Weeks 2, 8, and 16
Population: Randomized participants with a Baseline and at least one post-baseline measurement; last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 37 | 40 | 37 | 42
percent change
  Week 2: number analyzed (Participants) | 37 | 39 | 37 | 42
  Week 2 | 1.7 (5.59) | -29.3 (5.45) | -46.0 (5.44) | -57.6 (5.24)
  Week 8 | -6.7 (7.51) | -35.5 (7.28) | -45.1 (7.32) | -73.1 (7.05)
  Week 16 | -9.7 (8.30) | -39.6 (8.04) | -48.0 (8.08) | -68.9 (7.79)
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 2; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -59.3, 95% CI 2-sided [-72.3 to -46.3], Standard Error of Mean 6.58
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 2; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -47.7, 95% CI 2-sided [-61.1 to -34.3], Standard Error of Mean 6.78
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 2; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -31.1, 95% CI 2-sided [-44.3 to -17.8], Standard Error of Mean 6.7
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 8; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -66.4, 95% CI 2-sided [-83.9 to -48.9], Standard Error of Mean 8.85
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 8; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -38.4, 95% CI 2-sided [-56.4 to -20.4], Standard Error of Mean 9.13
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 8; Test type: Superiority; p = 0.002, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -28.9, 95% CI 2-sided [-46.6 to -11.2], Standard Error of Mean 8.96
Statistical Analysis 7: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 16; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -59.2, 95% CI 2-sided [-78.6 to -39.9], Standard Error of Mean 9.78
Statistical Analysis 8: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 16; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -38.3, 95% CI 2-sided [-58.3 to -18.4], Standard Error of Mean 10.08
Statistical Analysis 9: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of Percent Change from Baseline in Pruritus NRS at Week 16; Test type: Superiority; p = 0.003, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -29.9, 95% CI 2-sided [-49.4 to -10.3], Standard Error of Mean 9.90

5. Secondary Outcome: Percent Change From Baseline in EASI Score at Week 8
Description: EASI is a tool used to measure the extent (area) and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the area score is recorded as the percentage of skin affected by eczema. For each region, the severity score is calculated as the sum of the intensity scores (scored as none [0], mild [1)] moderate [2], or severe [3]) for Redness (erythema, inflammation), Thickness (induration, papulation, swelling - acute eczema), Scratching (excoriation), and Lichenification (lined skin, prurigo nodules - chronic eczema).
  The total EASI score for each region is calculated by multiplying the severity score by the area score, with adjustment for the proportion of the body region to the whole body. The final EASI score is the sum of the 4 region scores and ranges from 0 to 72 where higher scores represent worse disease; a negative change from Baseline indicates improvement.
Time Frame: Baseline and Week 8
Population: Randomized participants with at least one post-baseline measurement; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 39 | 42 | 42 | 42
percent change | -17.5 (6.27) | -43.7 (6.09) | -65.4 (5.97) | -82.8 (5.98)
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -65.3, 95% CI 2-sided [-80.0 to -50.5], Standard Error of Mean 7.46
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -47.9, 95% CI 2-sided [-62.6 to -33.3], Standard Error of Mean 7.42
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -26.2, 95% CI 2-sided [-40.8 to -11.5], Standard Error of Mean 7.42

6. Secondary Outcome: Percent Change From Baseline in SCORing Atopic Dermatitis (SCORAD) Score at Weeks 8 and 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline and Weeks 8 and 16
Population: Randomized participants with Baseline and at least one post-baseline measurement; Last observation carried forward imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 33 | 39 | 36 | 40
percent change
  Week 8 | -7.0 (5.84) | -35.4 (5.53) | -44.1 (5.69) | -65.3 (5.52)
  Week 16 | -12.4 (5.97) | -32.5 (5.66) | -46.9 (5.82) | -60.4 (5.65)
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of Percent Change from Baseline in SCORAD at Week 8; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -58.3, 95% CI 2-sided [-71.7 to -44.9], Standard Error of Mean 6.78
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of Percent Change from Baseline in SCORAD at Week 8; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -37.1, 95% CI 2-sided [-50.8 to -23.4], Standard Error of Mean 6.94
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of Percent Change from Baseline in SCORAD at Week 8; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -28.4, 95% CI 2-sided [-41.9 to -15.0], Standard Error of Mean 6.81
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of Percent Change from Baseline in SCORAD at Week 16; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -48.0, 95% CI 2-sided [-61.7 to -34.3], Standard Error of Mean 6.93
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of Percent Change from Baseline in SCORAD at Week 16; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -34.5, 95% CI 2-sided [-48.5 to -20.5], Standard Error of Mean 7.10
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of Percent Change from Baseline in SCORAD at Week 16; Test type: Superiority; p = 0.004, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -20.2, 95% CI 2-sided [-33.9 to -6.4], Standard Error of Mean 6.96

7. Secondary Outcome: Percentage of Participants Who Achieved an EASI 75 Response at Week 8
Description: EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  An EASI 75 response is defined as participants with at least a 75% reduction (improvement) in EASI score relative to the Baseline value.
  Participants with missing values at Week 8 were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Week 8
Population: All randomized participants; Non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants | 7.3 | 31.0 | 52.4 | 81.0
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 72.7, 95% CI 2-sided [58.3 to 87.1]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 44.9, 95% CI 2-sided [27.9 to 61.9]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.004, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 23.4, 95% CI 2-sided [7.5 to 39.4]

8. Secondary Outcome: Percentage of Participants Who Achieved an EASI 50 Response at Weeks 8 and 16
Description: EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  An EASI 50 response is defined as participants with at least a 50% reduction (improvement) in EASI score relative to the Baseline value.
  Participants with missing values at each time point were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Weeks 8 and 16
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants
  Week 8 | 22.0 | 54.8 | 71.4 | 92.9
  Week 16 | 22.0 | 50.0 | 71.4 | 83.3
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of EASI 50 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 70.7, 95% CI 2-sided [56.2 to 85.2]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of EASI 50 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 49.0, 95% CI 2-sided [30.8 to 67.3]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of EASI 50 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 32.8, 95% CI 2-sided [13.4 to 52.2]
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of EASI 50 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 60.6, 95% CI 2-sided [45.3 to 75.9]
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of EASI 50 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 48.6, 95% CI 2-sided [31.3 to 65.9]
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of EASI 50 Response at Week 16; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 28.2, 95% CI 2-sided [9.8 to 46.6]

9. Secondary Outcome: Percentage of Participants Who Achieved an EASI 90 Response at Weeks 8 and 16
Description: EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  An EASI 90 response is defined as participants with at least a 90% reduction (improvement) in EASI score relative to the Baseline value.
  Participants with missing values at each time point were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Weeks 8 and 16
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants
  Week 8 | 0.0 | 9.5 | 26.2 | 45.2
  Week 16 | 2.4 | 14.3 | 26.2 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of EASI 90 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 43.8, 95% CI 2-sided [29.1 to 58.5]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of EASI 90 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 26.1, 95% CI 2-sided [12.6 to 39.6]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of EASI 90 Response at Week 8; Test type: Superiority; p = 0.051, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 9.4, 95% CI 2-sided [-0.0 to 18.8]
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of EASI 90 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 46.9, 95% CI 2-sided [31.3 to 62.4]
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of EASI 90 Response at Week 16; Test type: Superiority; p = 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 23.8, 95% CI 2-sided [9.6 to 38.1]
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of EASI 90 Response at Week 16; Test type: Superiority; p = 0.049, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 11.8, 95% CI 2-sided [0.1 to 23.6]

10. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 50 Response at Weeks 8 and 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).
  A SCORAD 50 response is defined as participants with at least a 50% reduction (improvement) in SCORAD score relative to the Baseline value.
  Participants with missing values were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Weeks 8 and 16
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants
  Week 8 | 7.3 | 33.3 | 42.9 | 76.2
  Week 16 | 7.3 | 28.6 | 42.9 | 61.9
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of SCORAD 50 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 68.4, 95% CI 2-sided [54.0 to 82.8]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of SCORAD 50 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 35.3, 95% CI 2-sided [18.5 to 52.2]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of SCORAD 50 Response at Week 8; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 25.7, 95% CI 2-sided [9.6 to 41.7]
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of SCORAD 50 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 54.5, 95% CI 2-sided [39.0 to 69.9]
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of SCORAD 50 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 35.8, 95% CI 2-sided [19.1 to 52.5]
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of SCORAD 50 Response at Week 16; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 21.2, 95% CI 2-sided [5.7 to 36.8]

11. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 75 Response at Weeks 8 and 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).
  A SCORAD 75 response is defined as participants with at least a 75% reduction (improvement) in SCORAD score relative to the Baseline value.
  Participants with missing values were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Weeks 8 and 16
Population: All randomized participants; Non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants
  Week 8 | 0.0 | 9.5 | 9.5 | 31.0
  Week 16 | 2.4 | 4.8 | 21.4 | 40.5
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of SCORAD 75 Response at Week 8; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 30.4, 95% CI 2-sided [16.2 to 44.6]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of SCORAD 75 Response at Week 8; Test type: Superiority; p = 0.052, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 9.4, 95% CI 2-sided [-0.1 to 18.9]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of SCORAD 75 Response at Week 8; Test type: Superiority; p = 0.048, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 9.3, 95% CI 2-sided [0.1 to 18.5]
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of SCORAD 75 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 37.7, 95% CI 2-sided [22.2 to 53.3]
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of SCORAD 75 Response at Week 16; Test type: Superiority; p = 0.006, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 19.0, 95% CI 2-sided [5.6 to 32.5]
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of SCORAD 75 Response at Week 16; Test type: Superiority; p = 0.581, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 2.4, 95% CI 2-sided [-6.0 to 10.8]

12. Secondary Outcome: Percentage of Participants Who Achieved a SCORAD 90 Response at Weeks 8 and 16
Description: SCORAD is a clinical tool used to assess the extent and severity of eczema (SCORing Atopic Dermatitis). The extent is assessed using the rule of 9 to calculate the affected area (A) as a percentage of the whole body (0-100%). The intensity part of the SCORAD (B) consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness, each graded on a scale from 0 (none) to 3 (severe), for a total score of 0 to 18. Subjective items (C) include daily pruritus and sleeplessness, each scored on a visual analogue scale (VAS) from 0 to 10 (total score 0-20). SCORAD is calculated as A/5 + 7B/2 + C, and ranges from 0 to 103 (worst).
  A SCORAD 90 response is defined as participants with at least a 90% reduction (improvement) in SCORAD score relative to the Baseline value.
  Participants with missing values were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Weeks 8 and 16
Population: All randomized participants; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 41 | 42 | 42 | 42
percentage of participants
  Week 8 | 0.0 | 4.8 | 2.4 | 14.3
  Week 16 | 0.0 | 2.4 | 9.5 | 23.8
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of SCORAD 90 Response at Week 8; Test type: Superiority; p = 0.012, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 14.2, 95% CI 2-sided [3.2 to 25.2]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of SCORAD 90 Response at Week 8; Test type: Superiority; p = 0.428, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 2.3, 95% CI 2-sided [-3.4 to 8.0]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of SCORAD 90 Response at Week 8; Test type: Superiority; p = 0.206, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 4.6, 95% CI 2-sided [-2.5 to 11.8]
Statistical Analysis 4: Comparison: Placebo vs Upadacitinib 30 mg; Analysis of SCORAD 90 Response at Week 16; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 23.3, 95% CI 2-sided [10.4 to 36.2]
Statistical Analysis 5: Comparison: Placebo vs Upadacitinib 15 mg; Analysis of SCORAD 90 Response at Week 16; Test type: Superiority; p = 0.048, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 9.4, 95% CI 2-sided [0.1 to 18.8]
Statistical Analysis 6: Comparison: Placebo vs Upadacitinib 7.5 mg; Analysis of SCORAD 90 Response at Week 16; Test type: Superiority; p = 0.426, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 2.4, 95% CI 2-sided [-3.4 to 8.1]

13. Secondary Outcome: Percent Change From Re-randomization (Week 16) in EASI Score in Period 2
Description: as for outcome 1
Time Frame: Re-randomization (Week 16) and Weeks 20, 24, 32, 40, 52, 64, 76, and 88
Population: Participants who were re-randomized at the entry of Period 2 (Week 16) with at least one post-Week 16 assessment; Last observation carried forward (LOCF) imputation was used.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Placebo / Placebo | Placebo / Upadacitinib 30 mg | Upadacitinib 7.5 mg / Placebo | Upadacitinib 7.5 mg / Upadacitinib 7.5 mg | Upadacitinib 15 mg / Placebo | Upadacitinib 15 mg / Upadacitinib 15 mg | Upadacitinib 30 mg / Placebo | Upadacitinib 30 mg / Upadacitinib 30 mg
Number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 18 | 14 | 19
percent change
  Week 20: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 16 | 13 | 18
  Week 20 | 50.7 (33.50) | 11.8 (30.59) | 186.0 (46.53) | 79.1 (48.42) | 582.3 (172.19) | 65.7 (178.24) | 791.5 (262.34) | -73.8 (215.54)
  Week 24: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 16 | 13 | 19
  Week 24 | 13.5 (17.13) | -67.5 (15.64) | 189.6 (44.17) | 59.0 (45.97) | 607.3 (169.49) | 72.6 (175.44) | 898.5 (248.78) | -69.6 (200.01)
  Week 32: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 16 | 14 | 19
  Week 32 | -2.3 (15.15) | -83.1 (13.83) | 181.5 (44.74) | 63.5 (46.56) | 613.3 (169.63) | 151.7 (175.59) | 771.5 (252.90) | -28.8 (210.78)
  Week 40: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 16 | 14 | 18
  Week 40 | -31.2 (18.16) | -92.0 (16.58) | 200.9 (41.58) | 77.6 (43.27) | 608.8 (169.95) | 154.1 (175.92) | 778.9 (344.45) | 140.6 (293.17)
  Week 52: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 18 | 14 | 18
  Week 52 | -29.8 (17.74) | -90.1 (16.20) | 189.1 (43.65) | 74.4 (45.42) | 613.8 (166.85) | 104.1 (164.05) | 799.5 (254.30) | -13.3 (216.44)
  Week 64: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 18 | 14 | 18
  Week 64 | -35.8 (17.34) | -91.4 (15.83) | 179.9 (44.91) | 71.8 (46.74) | 614.6 (166.57) | 104.1 (163.78) | 802.1 (278.76) | 63.6 (237.26)
  Week 76: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 17 | 14 | 19
  Week 76 | -37.3 (19.09) | -90.3 (17.43) | 201.4 (41.89) | 77.7 (43.60) | 614.0 (168.03) | 130.2 (169.29) | 787.8 (262.89) | 24.4 (219.11)
  Week 88: number analyzed (Participants) | 10 | 10 | 15 | 15 | 17 | 18 | 14 | 18
  Week 88 | -37.7 (19.18) | -84.6 (17.51) | 170.7 (46.87) | 69.1 (48.78) | 617.5 (165.84) | 99.3 (163.06) | 769.7 (265.64) | 39.0 (226.10)

14. Secondary Outcome: Time to Loss of EASI 50 Response Relative to Baseline Among Participants Re-randomized as EASI 75 Responders at Week 16
Description: Time to loss of EASI 50 response in Period 2 relative to Baseline among those who were re-randomized as EASI 75 responders at Week 16.
  Time to loss of EASI 50 response was measured from Week 16 to the date of the first assessment in Period 2 where a participant's EASI score was higher than 50% of their Baseline score.
  Participants with no loss of response were censored at their last treatment visit or the start of rescue treatment, whichever occurred first.
Time Frame: From re-randomization at Week 16 until Week 88
Population: Participants who were re-randomized as EASI 75 responders at Week 16.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo / Placebo | Placebo / Upadacitinib 30 mg | Upadacitinib 7.5 mg / Placebo | Upadacitinib 7.5 mg / Upadacitinib 7.5 mg | Upadacitinib 15 mg / Placebo | Upadacitinib 15 mg / Upadacitinib 15 mg | Upadacitinib 30 mg / Placebo | Upadacitinib 30 mg / Upadacitinib 30 mg
Number analyzed (Participants) | 1 | 2 | 5 | 5 | 12 | 10 | 14 | 15
days | NA [NA to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events | 29 [27 to NA] — Could not be estimated due to the low number of events | NA [29 to NA] — Could not be estimated due to the low number of events | 30 [17 to 55] | 114 [29 to NA] — Could not be estimated due to the low number of events | 28 [25 to 36] | NA [NA to NA] — Could not be estimated due to the low number of events

15. Secondary Outcome: Percentage of Participants With an EASI 75 Response in Period 2 in Participants Who Were Re-randomized as EASI 75 Non-responders at Week 16
Description: EASI is a tool to measure the extent and severity of atopic eczema based on assessments of the head/neck, trunk, upper limbs and lower limbs. For each region the percentage of skin affected, and the severity of eczema (scored as none [0], mild [1], moderate [2], or severe [3]) for redness, thickness, scratching, and lichenification are assessed. The EASI score is the sum of the scores for each region and ranges from 0 to 72, where higher scores represent worse disease.
  An EASI 75 response is defined as at least a 75% reduction (improvement) in EASI score relative to the Baseline value, and was analyzed in participants who were re-randomized at Week 16 and were EASI 75 non-responders at Week 16.
Time Frame: Weeks 20, 24, 32, 40, 52, 64, 76, and 88
Population: Participants who were re-randomized at Week 16 and were EASI 75 non-responders at Week 16, and with available data at each time point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo / Placebo | Placebo / Upadacitinib 30 mg | Upadacitinib 7.5 mg / Placebo | Upadacitinib 7.5 mg / Upadacitinib 7.5 mg | Upadacitinib 15 mg / Placebo | Upadacitinib 15 mg / Upadacitinib 15 mg | Upadacitinib 30 mg / Placebo | Upadacitinib 30 mg / Upadacitinib 30 mg
Number analyzed (Participants) | 9 | 8 | 10 | 11 | 7 | 8 | 5 | 4
percentage of participants
  Week 20 | 11.1 | 12.5 | 0 | 9.1 | 0 | 12.5 | 20.0 | 25.0
  Week 24: number analyzed (Participants) | 1 | 7 | 0 | 3 | 1 | 2 | 3 | 3
  Week 24 | 100 | 85.7 |  | 33.3 | 0 | 0 | 33.3 | 33.3
  Week 32: number analyzed (Participants) | 1 | 6 | 0 | 2 | 1 | 2 | 2 | 2
  Week 32 | 100 | 100 |  | 0 | 0 | 50.0 | 50.0 | 50.0
  Week 40: number analyzed (Participants) | 1 | 6 | 0 | 0 | 1 | 1 | 1 | 2
  Week 40 | 100 | 66.7 |  |  | 0 | 100 | 0 | 50.0
  Week 52: number analyzed (Participants) | 1 | 6 | 0 | 0 | 1 | 1 | 0 | 2
  Week 52 | 100 | 66.7 |  |  | 0 | 100 |  | 50.0
  Week 64: number analyzed (Participants) | 1 | 5 | 0 | 0 | 1 | 1 | 0 | 1
  Week 64 | 100 | 80.0 |  |  | 0 | 100 |  | 100
  Week 76: number analyzed (Participants) | 1 | 3 | 0 | 0 | 1 | 1 | 0 | 1
  Week 76 | 100 | 100 |  |  | 0 | 100 |  | 100
  Week 88: number analyzed (Participants) | 1 | 2 | 0 | 0 | 1 | 1 | 0 | 1
  Week 88 | 100 | 100 |  |  | 0 | 100 |  | 100

16. Secondary Outcome: Percentage of Participants Who Achieved a Dermatology Life Quality Index (DLQI) of "0" or "1" at Weeks 8 and 16
Description: The DLQI is a 10-item questionnaire that asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week in the following 6 aspects: symptoms and feelings, daily activities, leisure, work or school activities, personal relationships and treatment related feelings. Participants answer the 10 questions on a scale from 0 (not at all) to 3 (very much). The DLQI is calculated by summing the scores of the 10 questions, resulting in a maximum of 30 and a minimum of 0 with higher scores indicating more impaired quality of life. A score of 0 or 1 means that the disease has no effect at all.
  Dermatology Life Quality Index outcomes were defined but are not reported because of an error in the programming of the electronic device used to administer the questionnaire that precluded determination of these outcomes.
Time Frame: Weeks 8 and 16
Population: Due to an error in the electronic device used to administer the questionnaire data were not available for any participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

17. Secondary Outcome: Change From Baseline in DLQI at Weeks 8 and 16
Description: The DLQI is a 10-item questionnaire that asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week in the following 6 aspects: symptoms and feelings, daily activities, leisure, work or school activities, personal relationships and treatment related feelings. Participants answer the 10 questions on a scale from 0 (not at all) to 3 (very much). The DLQI is calculated by summing the scores of the 10 questions, resulting in a maximum of 30 and a minimum of 0 with higher scores indicating more impaired quality of life. A negative change from Baseline indicates improvement.
  Dermatology Life Quality Index outcomes were defined but are not reported because of an error in the programming of the electronic device used to administer the questionnaire that precluded determination of these outcomes.
Time Frame: Baseline and Weeks 8 and 16
Population: as for outcome 16
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Percentage of Body Surface Area (BSA) Affected by Atopic Dermatitis at Week 16
Description: Body surface area (BSA) affected by atopic dermatitis was assessed by the physician and is expressed as a percentage of the total BSA. For purposes of the estimation, the total surface of the participant's palm plus five digits was assumed to be approximately equivalent to 1% BSA.
  Last observation carried forward imputation was used.
Time Frame: Baseline and Week 16
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 39 | 42 | 42 | 42
percentage of body surface area | -4.1 (3.58) | -11.7 (3.48) | -27.1 (3.43) | -30.7 (3.43)
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -26.5, 95% CI 2-sided [-34.9 to -18.1], Standard Error of Mean 4.25
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -23.0, 95% CI 2-sided [-31.4 to -14.6], Standard Error of Mean 4.27
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.075, ANCOVA; ANCOVA with stratum (geographic region), baseline value, and treatment in the model; LS Mean Difference = -7.6, 95% CI 2-sided [-16.0 to 0.8], Standard Error of Mean 4.25

19. Secondary Outcome: Percentage of Participants With Reduction of ≥ 4 Points From Baseline in Pruritus NRS at Week 16
Description: Participants were asked to rate pruritus (itch) in the past 24 hours on a daily basis using a scale from 0 to 10, with 0 being no itch and 10 being the worst imaginable itch. The percentage of participants with reduction of ≥ 4 points from Baseline in pruritus NRS was assessed in participants with a baseline pruritus NRS of ≥ 4. Participants with missing values at Week 16 were counted as non-responders in this analysis (non-responder imputation).
Time Frame: Baseline and Week 16
Population: Randomized participants with Baseline pruritus NRS of ≥ 4; non-responder imputation was used.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Upadacitinib 7.5 mg | Upadacitinib 15 mg | Upadacitinib 30 mg
Number analyzed (Participants) | 35 | 37 | 32 | 36
percentage of participants | 5.7 | 24.3 | 59.4 | 52.8
Statistical Analysis 1: Comparison: Placebo vs Upadacitinib 30 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 47.4, 95% CI 2-sided [29.6 to 65.2]
Statistical Analysis 2: Comparison: Placebo vs Upadacitinib 15 mg; Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 53.4, 95% CI 2-sided [35.5 to 71.3]
Statistical Analysis 3: Comparison: Placebo vs Upadacitinib 7.5 mg; Test type: Superiority; p = 0.021, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratum (geographic region); Adjusted Difference = 18.6, 95% CI 2-sided [2.8 to 34.3]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug up to 30 days after last dose. Period 1: 16 weeks, Period 2: 72 weeks.
Description: Any adverse event that occurred on or after the first dose of upadacitinib 30 mg rescue therapy in Period 2 is counted in the Period 1+2: Upadacitinib 30 mg group. Participants who received rescue therapy after placebo, upadacitinib 7.5 mg or 15 mg treatment in Period 2 are counted in the denominators of both Period 1+2: Placebo/Upadacitinib 7.5 mg/15 mg and Period 1+2: Upadacitinib 30 mg dose groups.
Groups:
- Period 1: Placebo: Participants received placebo once daily (QD) for 16 weeks in Period 1.
- Period 1: Upadacitinib 7.5 mg: Participants received upadacitinib 7.5 mg once daily for 16 weeks in Period 1
- Period 1: Upadacitinib 15 mg: Participants received upadacitinib 15 mg once daily for 16 weeks in Period 1.
- Period 1: Upadacitinib 30 mg: Participants received upadacitinib 30 mg once daily for 16 weeks in Period 1.
- Period 1+2: Upadacitinib 7.5 mg: Participants originally randomized to upadacitinib 7.5 mg received upadacitinib 7.5 mg once daily for 16 weeks in Period 1; Participants re-randomized to upadacitinib 7.5 mg in Period 2 continued to receive upadacitinib 7.5 mg for 72 weeks in Period 2 or until rescue.
- Period 1+2: Upadacitinib 15 mg: Participants originally randomized to upadacitinib 15 mg received upadacitinib 15 mg once daily for 16 weeks in Period 1; Participants re-randomized to upadacitinib 15 mg in Period 2 continued to receive upadacitinib 15 mg for 72 weeks in Period 2 or until rescue.
- Period 1+2: Upadacitinib 30 mg: Participants originally randomized to upadacitinib 30 mg received upadacitinib 30 mg once daily for 16 weeks in Period 1. Participants re-randomized to upadacitinib 30 mg in Period 2 continued to receive upadacitinib 30 mg for 72 weeks in Period 2.
  Participants originally randomized to placebo and re-randomized to upadacitinib 30 mg at Week 16 received upadacitinib 30 mg from Week 16 to Week 88.
  Participants re-randomized to placebo, upadacitinib 7.5 mg or 15 mg at Week 16 who were rescued starting at Week 20 or later received upadacitinib 30 mg until Week 88.
- Period 1+2: Placebo: Participants originally randomized to placebo received placebo once daily for 16 weeks in Period 1.
  Participants re-randomized to placebo in Period 2 continued to receive placebo for 72 weeks in Period 2 or until rescue.
Arm/Group | Period 1: Placebo | Period 1: Upadacitinib 7.5 mg | Period 1: Upadacitinib 15 mg | Period 1: Upadacitinib 30 mg | Period 1+2: Upadacitinib 7.5 mg | Period 1+2: Upadacitinib 15 mg | Period 1+2: Upadacitinib 30 mg | Period 1+2: Placebo
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/42 | 0/42 | 0/42 | 0/42 | 0/42 | 2/114 | 0/93
Serious Adverse Events (participants affected / at risk) | 1/40 | 2/42 | 1/42 | 0/42 | 2/42 | 1/42 | 7/114 | 1/93
Other Adverse Events (participants affected / at risk) | 15/40 | 21/42 | 17/42 | 21/42 | 23/42 | 22/42 | 68/114 | 19/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=40) | Period 1: Upadacitinib 7.5 mg (N=42) | Period 1: Upadacitinib 15 mg (N=42) | Period 1: Upadacitinib 30 mg (N=42) | Period 1+2: Upadacitinib 7.5 mg (N=42) | Period 1+2: Upadacitinib 15 mg (N=42) | Period 1+2: Upadacitinib 30 mg (N=114) | Period 1+2: Placebo (N=93)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OESOPHAGEAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERICORONITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: Placebo (N=40) | Period 1: Upadacitinib 7.5 mg (N=42) | Period 1: Upadacitinib 15 mg (N=42) | Period 1: Upadacitinib 30 mg (N=42) | Period 1+2: Upadacitinib 7.5 mg (N=42) | Period 1+2: Upadacitinib 15 mg (N=42) | Period 1+2: Upadacitinib 30 mg (N=114) | Period 1+2: Placebo (N=93)
DIARRHOEA (Gastrointestinal disorders) | 2 (2) | 2 (2) | 2 (4) | 0 (0) | 2 (2) | 2 (5) | 2 (2) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 6 (8) | 2 (2)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 10 (10) | 0 (0)
IMPETIGO (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 8 (8) | 0 (0)
INFLUENZA (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 2 (2) | 4 (5) | 3 (3) | 3 (3) | 5 (6) | 11 (16) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (4) | 7 (7) | 5 (5) | 5 (9) | 7 (7) | 7 (7) | 26 (47) | 5 (5)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 6 (8) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 2 (2) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 3 (3) | 7 (8) | 3 (3)
HEADACHE (Nervous system disorders) | 1 (1) | 3 (3) | 3 (3) | 4 (4) | 3 (3) | 3 (3) | 7 (7) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PROTEINURIA (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 2 (2) | 6 (7) | 4 (6) | 2 (2) | 13 (14) | 1 (1)
DERMATITIS ATOPIC (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (6) | 2 (2) | 4 (5) | 6 (7) | 5 (5) | 22 (25) | 2 (2)
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2017-08-30): https://cdn.clinicaltrials.gov/large-docs/17/NCT02925117/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/17/NCT02925117/SAP_001.pdf